CLINICAL TRIAL: NCT02065115
Title: Cryoanalgesia (Ice Pack) to Reduce the Pain Associated With Arterial Blood Gas Puncture
Brief Title: Study of Ice Application to Reduce Pain From Arterial Punctures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph Hospital, New Hampshire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SJH IRB 2012-05
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Vessel Puncture Site Pain
Keywords: ice; cryotherapy; puncture; pain
MeSH Terms: conditions — Pain | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cryotherapy (Experimental): Cryotherapy: 12 ounces of crushed ice place in a plastic bag applied to the radial artery puncture area for 3 minutes
  Interventions: Other: Cryotherapy (ice pack)
- Control (No Intervention): Cryotherapy is not applied to the radial artery puncture area

INTERVENTIONS:
Other: Cryotherapy (ice pack)
  Arms: Cryotherapy

SUMMARY:
This study seeks to determine if cryoanalgesia in the form of ice application could be an effective analgesic when applied before arterial puncture.

ELIGIBILITY:
Inclusion Criteria:

* subjects ≥ 18 years old referred to the pulmonary function laboratory with a physician order for an arterial blood gas test were sought to complete the study

Exclusion Criteria:

* cold, bluish hands and fingers
* diagnosis of Raynaud's syndrome or scleroderma/CREST syndrome
* history or signs of dementia, confusion, or cognitive impairment
* blindness
* patients not fluent in the English language
* non-palpable radial pulse in the wrist (necessitating brachial puncture)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
pain related to arterial puncture | 1-5 minutes after arterial puncture
  Pain is measured with a 100 mm visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey m Haynes, RRT RPFT, Principal Investigator — St. Joseph Hospital, Nashua New Hampshire
Locations (1):
- St. Joseph Hospital, Nashua, New Hampshire, United States

REFERENCES:
- [Background] Giner J, Casan P, Belda J, Gonzalez M, Miralda RM, Sanchis J. Pain during arterial puncture. Chest. 1996 Dec;110(6):1443-5. doi: 10.1378/chest.110.6.1443. PMID 8989058
- [Derived] Haynes JM. Randomized controlled trial of cryoanalgesia (ice bag) to reduce pain associated with arterial puncture. Respir Care. 2015 Jan;60(1):1-5. doi: 10.4187/respcare.03312. Epub 2014 Dec 16. PMID 25516991